CLINICAL TRIAL: NCT01210209
Title: GENEWING - A Genome Wide Association Study in Ewing Sarcoma
Brief Title: Study of Blood Samples From Patients With Ewing Sarcoma and Their Relatives
Acronym: GENEWING
Status: Completed | Type: Observational
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Other Study IDs: IC 2009-02; CLCC-IC-2009-02; 2009-A00558-49; EU-21064
Record Dates: First submitted 2010-09-25; First posted 2010-09-28 (Estimated); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Sarcoma
Keywords: Ewing sarcoma; Ewing sarcoma/peripheral primitive neuroectodermal tumor (PNET)
MeSH Terms: conditions — Sarcoma; Sarcoma, Ewing; Neuroectodermal Tumors, Primitive, Peripheral | interventions — Genome-Wide Association Study

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: genome-wide association study

SUMMARY:
RATIONALE: Studying samples of blood in the laboratory from patients with cancer and their relatives may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is looking at blood samples collected from patients with Ewing sarcoma and their relatives.

DETAILED DESCRIPTION:
OBJECTIVES:

* To identify and characterize a genetic susceptibility factor to Ewing's sarcoma by performing a Genome-Wide Association Study with as many as possible Ewing sarcoma patients.

OUTLINE: This is a multicenter study.

Blood samples are collected from patients and their relatives. Blood DNA samples are analyzed for susceptibility genes of Ewing Sarcoma.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients with Ewing sarcoma
* Relatives of Ewing sarcoma patients

PATIENT CHARACTERISTICS:

* Patients with a fusion genes specific of Ewing Sarcoma

PRIOR CONCURRENT THERAPY:

* Not applicable

Ages: 0 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Ewing's sarcoma, with idenfication of a specific translocation of Ewing's sarcoma
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2010-01-07 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Identification and characterization of susceptibility genes in patients with Ewing sarcoma | Through study completion, an average of 10 years
  Identification and characterization of susceptibility genes in patients with Ewing sarcoma

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Delattre, MD, Principal Investigator — Institut Curie
Locations (1):
- Institut Curie Hopital, Paris, France

REFERENCES:
- See also: InCa — http://www.e-cancer.fr/Professionnels-de-sante/Le-registre-des-essais-cliniques/Le-registre-des-essais-cliniques/Etudes-cliniques/GENEWING-Essai-visant-a-identifier-et-caracteriser-des-genes-de-susceptibilite-au-sarcome-d-Ewing-chez-des-patients-ayant-un-sarcome-d-Ewing-et-leurs-proches-parents.-essai-clos-aux-inclusions